CLINICAL TRIAL: NCT02011100
Title: Randomised Placebo Controlled Study of the Effect of Carnosine Diabetes and Cardiovascular Risk Factors
Brief Title: Effect of Carnosine on Diabetes and Cardiovascular Risk Factors
Acronym: Carnorisk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jozef Ukropec (Other Government)
Responsible Party: Sponsor-Investigator, Jozef Ukropec, PhD, Slovak Academy of Sciences
Organization: Slovak Academy of Sciences (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CarnoDMCVD
Record Dates: First submitted 2013-12-05; First posted 2013-12-13 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Metabolic Diseases, Type 2 Diabetes, Cardiovascular Disease
MeSH Terms: conditions — Metabolic Diseases; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Carnosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CARNOSINE (Experimental): 3 months oral carnosine administration in a dose of 2 gram per day, twice a day 1 gram dose (1-0-1)
  Interventions: Dietary Supplement: Carnosine
- placebo (Placebo Comparator): 3 months placebo intake - taken twice a day (1-0-1)
  Interventions: Dietary Supplement: Carnosine

INTERVENTIONS:
Dietary Supplement: Carnosine

SUMMARY:
Carnosine is a naturally occurring compound with a potential health benefits. In animal studies, carnosine supplementation reduces manifestation of chronic civilization diseases, regulates subclinical inflammation, protein glycation and lipid & glucose metabolism. Our preliminary data showed the relationship between insulin resistance and carnosine content in human skeletal muscle. Based on these unique results we plan to perform intervention study aimed at identifying effects of carnosine on insulin sensitivity and secretion, which might reduce the development of T2D in obese. Similar metabolic effects of vitamin D3 were associated with expression of specific miRNAs. Circulating miRNAs related to carnosine action are unknown. The putative positive effects of carnosine on insulin sensitivity and secretion in obese patients might have a tremendous impact in prevention of type 2 diabetes. Identification of miRNAs associated with carnosine action could provide predictors of successful therapy.

ELIGIBILITY:
Inclusion Criteria:

* BMI (28-38 kg.m-2);
* waist circumference >94 cm;
* % body fat 30%
* fasting glycemia < 7 mmol/l

Exclusion Criteria:

* age < 25 or > 50 years,
* change in body weight > 5 kg in last 12 months,
* obesity with BMI > 38kg.m-2,
* previously or newly (oGTT) diagnosed type 2 diabetes,
* allergy, smoking, alcohol abuse, any pharmacotherapy including regular vitamin intake;
* cardiovascular, hematologic, respiratory, gastrointestinal, endocrine or oncologic diseases,
* kidney disease, acute inflammatory disease.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-12; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
oxidative stress | within one year
  AGEs and lipid peroxidation products
chronic systemic inflammation | one year
  circulating hsCRP

SECONDARY OUTCOMES:
level of glucose intolerance | within 10 months
  detected by the oral glucose tolerance test. expressed as 2h glucose, area under the glycemic curve, QUICKI index, HOMA-IR

OTHER OUTCOMES:
muscle carnosine content | within 9 months
  assessed by 1H-MRS of muscle in vivo (7T Magnet, Siemens, Germany) it will be expressed relative to creatine signal.

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Ukropec, PhD, Principal Investigator — Institute of experimental endocrinology SAS; Barbara Ukropcova, MD, PhD, Study Director — Faculty of Medicine Comenius University & Institute of Experimental Endocrinology SAS; Boris Krahulec, MD, PhD, Study Chair — University Hospital in Bratislava; Barbora deCourten, MD, MPH, PhD, FRACP, Study Chair — Monash University
Locations (2):
- Slovakia (2):
  - Univeristy Hospital in Bratislava, Bratislava
  - Institute of Experimental Endocrinology Slovak Academy of Sciences, Bratislava